CLINICAL TRIAL: NCT02500641
Title: The Effect of Intensive Urate Lowering Therapy (ULT) With Febuxostat in Comparison With Allopurinol on Cardiovascular Risk in Patients With Gout Using Surrogate Markers: a Randomized, Controlled Trial
Brief Title: Intensive Urate Lowering Therapy of Febuxostat Compared to Allopurinol on Cardiovascular Risk in Patients With Gout
Acronym: FORWARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini International Operations Luxembourg SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEIN/14/FEB-PWV/001; 2014-005567-33 (EudraCT Number)
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Gout
Keywords: Biological Markers; Cardiovascular disease; Humans; Pulse Wave Velocity; Cardiovascular risk factors; Allopurinol; Pulse Wave Analysis; Thiazoles; Inflammation; Uric acid; Febuxostat; Oxidative stress; Tumor Necrosis Factor; Arthritis; Hyperuricemia
MeSH Terms: conditions — Gout; Cardiovascular Diseases; Inflammation; Arthritis; Hyperuricemia | interventions — Febuxostat; Allopurinol; Colchicine; Naproxen; Omeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study physician, responsible for randomization and drug supply handling, was unblinded to study medications and therefore not involved in the main efficacy evaluations of each patient randomized in the study.
  Conversely, the study physician/s responsible for the main efficacy evaluation (Pulse Wave Velocity) was blinded to study treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Febuxostat 80/120 mg/day (Experimental): Febuxostat 80/120 mg film coated tablets.The initial daily dose is 80 mg given orally. In case a patient has serum urate level 6 mg/dl after 2 weeks of treatment the dose will be escalated to 120 mg and if tolerated will be maintained during the study treatment period.
  To prevent flares in the initial stages of treatment, patients will be treated for at least 6 months with colchicine 0.5 - 1 mg quaque die (QD ) or in case of colchicine intolerance, Naproxen 550 mg bis in die (BID) with Omeprazole (20-40 mg once daily), if indicated to be used.
  Interventions: Drug: Febuxostat 80/120mg/day; Drug: Colchicine; Drug: Naproxen; Drug: Omeprazole
- Allopurinol 100 up to 600 mg/day (Active Comparator): Allopurinol 100/300 mg tablets.The initial daily allopurinol dose is 100 mg given orally, to be escalated of 100 mg every 2 weeks in patients with serum urate concentration >6 mg/dl.
  The maximum dose of allopurinol achievable in the study will depend on kidney function and tolerability, but will not exceed 600 mg daily.To prevent flares in the initial stages of treatment, patients will be treated for at least 6 months with colchicine 0.5 - 1 mg QD or in case of colchicine intolerance, Naproxen 550 mg BID with Omeprazole (20-40 mg once daily), if indicated to be used.
  Interventions: Drug: Allopurinol 100 up to 600mg/day; Drug: Colchicine; Drug: Naproxen; Drug: Omeprazole

INTERVENTIONS:
Drug: Febuxostat 80/120mg/day — Starting dose and dose regimen of Febuxostat : the initial daily dose is 80 mg. In case the patient has the serum urate concentration > 6 mg/dl after 2 weeks of treatment the dose will be escalated to 120 mg and if tolerated will be maintained for the duration of the study.
  Other Names: Adenuric
  Arms: Febuxostat 80/120 mg/day
Drug: Allopurinol 100 up to 600mg/day — Starting dose and dose regimen of allopurinol : the initial daily allopurinol dose is 100 mg, to be increased by 100 mg every 2 weeks in patients with serum urate concentration >6 mg/dl. The maximum daily dose of allopurinol achievable in the study will depend on kidney function and tolerability, but will not exceed 600 mg.
  Other Names: Allopurinol
  Arms: Allopurinol 100 up to 600 mg/day
Drug: Colchicine — Colchicine 0.5 mg tablets.To prevent flares in the initial stages of treatment, patients will be treated for at least 6 months with colchicine 0.5 - 1 mg QD
Drug: Naproxen — Naproxen sodium 550 mg film coated tablets. In case of colchicine intolerance patients will be treated for at least 6 months with Naproxen 550 mg BID and Omeprazole (20-40 mg once daily), if indicated to be used.
  Other Names: Synflex
Drug: Omeprazole — Omeprazole 20 mg capsules, co-administered to patients for gastric protection.
  Other Names: Omeprazen

SUMMARY:
There is a mounting and clear association between hyperuricaemia, gout and the presence of traditional cardiovascular (CV) risk factors and CV event-equivalent conditions such as chronic kidney disease, metabolic syndrome, and diabetes. Gout is associated with increased risk of CV events such as myocardial infarction and CV death. Furthermore hyperuricaemia is clearly associated with an increased arterial stiffness, a marker of pre-clinical atherosclerosis. Carotid-femoral pulse wave velocity (PWV) is the "gold standard" measurement of arterial stiffness and it is considered, in this trial, as a valid surrogate endpoint with clearly established relevance to predict cardiovascular disease (CVD) clinical outcome In this randomised trial conducted on adult subjects with a history of gout, we use surrogate endpoints to investigate the efficacy of febuxostat compared with allopurinol to predict (CVD) clinical outcome.

Eligible subjects were randomised in a 1:1 ratio to the following treatment groups:

* Test product: febuxostat 80 mg or 120 mg once daily (120 mg daily, if serum urate was >6 mg/dL after 2 weeks of treatment at 80 mg daily).
* Active comparator: allopurinol 100 mg once daily (up to a maximum dose of 600 mg daily escalated in 100 mg increments every 2 weeks, if serum urate acid (sUA) was >6 mg/dL after 2 weeks of treatment at the previous dose).

The study duration was 39 weeks, which included the:

* Run-in/screening period: 1 week (extendable up to a maximum of 30 days according to variability of sUA levels);
* Treatment period: 36 weeks;
* Safety follow-up period: 2 weeks.

DETAILED DESCRIPTION:
The study physician, responsible for randomization and drug supply handling, is unblinded to study medications and therefore will not be involved in the main efficacy evaluations of each patient randomized in the study.

Conversely, the study physician/s responsible for the main efficacy evaluation (Pulse Wave Velocity) will be blind to study treatments.

Key efficacy variables will be performed by an independent centralized laboratory.

Trial was conducted in a detailed and orderly manner in accordance with established research principles, International Conference on Harmonization (ICH), Good Clinical Practice (GCP) Guidelines and with Clinical Research Organization (CRO) Standard Operating Procedures (SOPs). As part of a concerted effort to fulfill these obligations, the authorised CRO study monitor visited investigative sites prior to and during the trial in addition to maintaining telephone and written communication. Data from each subject were reviewed and source verified as the study progressed.

In accordance with audit plans, this trial may have been selected for audits. The investigators committed to permit independent audits by auditors assigned by the Sponsor at a reasonable notice. Audits included, but were not limited to, drug supply, presence of required documents, the informed consent process, protection of rights and well-being of subjects and verification of Electronic case report form (eCRF) entries against source documents.

Regulatory authorities worldwide had the right to inspect the investigative sites during or after the trial. In such cases, the investigators were required to contact the Sponsor immediately and to fully cooperate with the inspectors.

Copies of written correspondence between the investigators, CRO, Sponsor, Competent Authorities, Institutional Review Board (IRB) and Independent Ethic Committee (IEC) are on file with the Sponsor and investigators.

Adverse events were according to the Medical Dictionary for Regulatory Activities (MedDRA, version 18.0) thesaurus.

Statistical analysis were conducted according the Statistical Analysis Plan (SAP) describing the analytical principles and statistical techniques employed in order to address the objectives specified in the Protocol.

A Data Management Plan was present for missing data, to address situations where variables are reported as missing, unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years and older;
2. History of gout, flare free in the 4 weeks prior to study entry
3. History of crystal (joint liquid) proven diagnosis or anamnestic diagnosis of gout according to Wallace at el. To be eligible, a subject had to present at least 6 of the following 12 clinical, laboratory, and x-ray phenomena:

1. Maximum inflammation developed within 1 day, 2. More than one attack of acute arthritis, 3. Monoarticular arthritis attack, 4. Redness observed over joints, 5. First metatarsophalangeal (MTP) pain or swelling, 6. Unilateral first MTP joint attack, 7. Unilateral tarsal joint attack, 8. Suspected or proven tophus, 9. Hyperuricemia, 10. Asymmetric swelling within a joint on a X ray, 11. Subcortical cysts without erosions on X ray, 12. Negative organisms on culture of joint fluid; 4. Naive to ULT or previously treated with ULT, but with no ULT treatment in the last 1 month prior to study entry and only if reason for ULT interruption was not due to safety concerns.

5. Patients at study entry have elevated serum urate level >8 mg/dl. 6. Overall Cardiovascular (CV) risk based on the scoring proposed by the Joint Task Force of the European Society of Cardiology and other European Societies on cardiovascular disease prevention in clinical practice between 5 and 15-% (inclusive). Patients with diabetes mellitus type 2 could be included in the study if their CV risk score is calculated as ≤7%.

7. Allowed concomitant medications should be maintained stable during the last 2 weeks before randomisation

Exclusion Criteria:

1. Severe chronic renal failure (creatinine clearance < 30 ml/min)
2. Hepatic failure
3. Active liver disease or hepatic dysfunction, defined as both alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2 times the upper limit of normal.
4. Diabetes mellitus type1
5. Life-threatening co-morbidity or with a significant medical condition and/or conditions that would interfere with the treatment, the safety or the compliance with the protocol
6. Diagnosis of, or receiving treatment for malignancy (excluding basalioma skin cancer) in the previous 5 years
7. Patients who have experienced either myocardial infarction or stroke
8. Patients with inflammatory based arthritis (e.g.: rheumatoid arthritis, etc.)
9. Patients with congestive heart failure, New York Heart Association (NYHA) Class III or IV
10. Patients with untreated/uncontrolled thyroid function
11. Patients with clinically severe peripheral arterial disease
12. Concomitant administration of any of the following: azathioprine, mercaptopurine, theophylline, meclofenamate, sulfinpyrazone, trimethoprim-sulfamethoxazole, cyclophosphamide, benzbromarone, pyrazinamide, captopril and enalapril (for Allopurinol), tegafur, pegloticase and tacrolimus.
13. Hypersensitivity to any one of the active substances or to any of the excipients
14. Any contraindication to febuxostat or allopurinol (with reference to the summary of product characteristics).
15. Subject is unable to take either of the protocol-required gout flare prophylactic medications (NSAID or colchicine) due to contraindications or intolerance, e.g. hypersensitivity, active gastric ulcer disease, renal impairment and/or changes in liver enzymes
16. Participation in another trial of an investigational drug or device within 30 days prior to screening, or prior treatment with investigational product(s)
17. Women of childbearing potential (WOCBP), including peri-menopausal women who have had a menstrual period within 1 year, not willing to use highly effective method of birth control throughout the study period and for 4 weeks after study completion defined as a method which results in a failure rate of less than 1% per year such as:

    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal),
    * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable),
    * intrauterine device (IUD),
    * intrauterine hormone-releasing system (IUS),
    * bilateral tubal occlusion,
    * vasectomised partner (provided that partner is the sole sexual partner of the trial participant and that the vasectomised partner has received medical assessment of the surgical success),
    * sexual abstinence;
18. Severe psychiatric disorders/neurological disorders
19. Severe concurrent pathology, including terminal illness (cancer, AIDS, etc)
20. Abuse of alcohol, analgesics, or psychotropic drugs
21. Inability or unwillingness, in the investigator's opinion, to follow study procedures including, but not limited to the ability to obtain adequate PWV/Pulse Wave Analysis (PWA) recordings. Special attention was made to any physical abnormalities which could affect quality of PWV/PWA measurement:

    * Neck region- neck flexibility and accessibility of carotid artery,
    * Upper arm and thigh region- exclude any abnormalities which would prevent adequate placement of the cuff;
22. Inability or unwillingness to issue the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, Prof, Study Director — Policlinico S.Orsola - Malpighi Medicina Interna Borghi
Locations (26):
- Medizinische Klinik und Poliklinik III/Rheumatologie Universitätsklinikum "Carl Gustav Carus" Der Technischen Universität, Dresden, Germany
- Italy (4):
  - Presidio Ospedaliero San Filippo e Nicola Università degli Studi dell'Aquila U.O.C Geriatria e Lungodegenza Geriatrica, Avezzano, L'Aquila
  - Ospedale San Salvatore U.O.C. Medicina Interna e Nefrologia Dipartimento MeSVA Università degli Studi dell'Aquila, Coppito, L'Aquila
  - Azienda Ospedaliero-Universitaria Policlinico Sant'Orsola-Malpighi, Bologna
  - Ospedale Policlinico SS. Annunziata Università degli Studi "G. d'Annunzio". Dipartimento di Medicina e Scienze dell'Invecchiamento., Chieti
- Reade Clinic, Amsterdam, Netherlands
- Poland (10):
  - Gdańskie Centrum Zdrowia Sp.z o.o., Gdansk
  - Specjalistyczna Praktyka Lekarska Piotr Kubalski, Grudziądz
  - Centrum Medyczne Pratia Katowice, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II w Krakowie, Krakow
  - Specjalistyczny Gabinet Dermatologiczno-Kosmetyczny, Krakow
  - Oddział Kardiologiczny, WSS im. W. Biegańskiego w Łodzi, Lodz
  - Polimedica, Lodz
  - Pratia S,A, Warsaw
  - Reumatika- Centrum Reumatologii, Warsaw
- Romania (6):
  - Clinica Medicală Data Plus SRL, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - S.C. Centrul Medical Sana S.R.L., Bucharest
  - S.C. Cardiomed S.R.L., Craiova
  - Cabinet Medical Medicina Interna, Timișoara
  - Institutul de Boli Cardiovasculare Clinica de Cardiologie si Recuperare Cardiovasculara, Timișoara
- Serbia (4):
  - Institut za kardiovaskularne bolesti Dedinje, Belgrade
  - Institut za reumatologiju, Belgrade
  - Kliničko-bolnički centar "Bežanijska kosa" Klinika za imunologiju i alergologiju, Belgrade
  - Vojnomedicinska akademija Klinika za reumatologiju, Belgrade

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A Run-in/screening period of 1 week (extendable up to a maximum of 30 days to account for variability of serum urate levels) was present prior than randomization.
Groups:
- Allopurinol 100 up to 600 mg/Day: Allopurinol 100/300 mg tablets.The initial daily allopurinol dose is 100 mg given orally, to be escalated of 100 mg every 2 weeks in patients with serum urate concentration >6 mg/dl.
  The maximum dose of allopurinol achievable in the study will depend on kidney function and tolerability, but will not exceed 600 mg daily.To prevent flares in the initial stages of treatment, patients will be treated for at least 6 months with colchicine 0.5 - 1 mg QD or in case of colchicine intolerance, Naproxen 550 mg BID with Omeprazole (20-40 mg once daily), if indicated to be used.
  Allopurinol 100 up to 600mg/day: Starting dose and dose regimen of allopurinol : the initial daily allopurinol dose is 100 mg, to be increased by 100 mg every 2 weeks in patients with serum urate concentration >6 mg/dl. The maximum daily dose of allopurinol achievable in the study will depend on kidney function and tolerability, but will not exceed 600 mg.
  Colchicine: Colchicine 0.5 mg tablets.To prevent flares in
Period: Overall Study
Arm/Group | Febuxostat 80/120 mg/Day | Allopurinol 100 up to 600 mg/Day
Started | 98 | 98
Completed | 88 | 86
Not Completed | 10 | 12
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Unable to follow study procedures | 3 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Sponsor decision | 1 | 0
Not completed — Non compliance to study drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomozed participants who had taken at least one dose of study drug specified by treatment group
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat 80/120 mg/Day | Allopurinol 100 up to 600 mg/Day | Total
Number analyzed (Participants) | 98 | 98 | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 60 | 128
  >=65 years | 30 | 38 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.66 (10.83) | 60.52 (10.35) | 59.59 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 81 | 80 | 161
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 1 | 0 | 1
  Romania | 27 | 25 | 52
  Poland | 38 | 52 | 90
  Italy | 9 | 6 | 15
  Serbia | 20 | 12 | 32
  Germany | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pulse Wave Velocity
Description: Comparison of the effects of Febuxostat and Allopurinol on Pulse Wave Velocity (PWV) after 36 weeks of treatment.
Time Frame: 36 weeks of treatment
Population: All randomized subjects who had taken at least one dose of study drug specified by treatment group and performed at least one primary efficacy assessment (PWV) after randomization.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Febuxostat 80/120 mg/Day | Allopurinol 100 up to 600 mg/Day
Number analyzed (Participants) | 92 | 90
m/s | 9.0 (2.04) | 9.05 (1.99)
Statistical Analysis 1: Comparison: Febuxostat 80/120 mg/Day vs Allopurinol 100 up to 600 mg/Day; Test type: Superiority; p = 0.5298, ANCOVA

ADVERSE EVENTS:
Time Frame: From signing of informed consent at visit -1 (from 7 to 30 days before treatment phase in case of retesting) to follow-up period of 2 weeks after the administration of the last treatment dose. Treatment duration was of 36 weeks.
Description: Adverse event's were considered abnormalities in laboratory analyses (newly occurring after administration or worsening of previously known abnormalities) considered clinically relevant by the Principal investigator (values significantly above or under normal range or requiring an intervention or diagnostic tests or may result in the Investigational Medical Product discontinuation).
Arm/Group | Febuxostat 80/120 mg/Day | Allopurinol 100 up to 600 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/98
Serious Adverse Events (participants affected / at risk) | 10/98 | 8/98
Other Adverse Events (participants affected / at risk) | 50/98 | 61/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Febuxostat 80/120 mg/Day (N=98) | Allopurinol 100 up to 600 mg/Day (N=98)
aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Adhesiolysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Large intestine operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Post Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ischemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Febuxostat 80/120 mg/Day (N=98) | Allopurinol 100 up to 600 mg/Day (N=98)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
edema peripheral (General disorders) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 0 (0)
Blood glucose increased (Investigations) | 3 (3) | 4 (4)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 0 (0)
Blood triglycerides increased (Investigations) | 2 (2) | 3 (3)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
eosinophil count decreased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 3 (3)
Heamoglobin decreased (Investigations) | 1 (1) | 2 (2)
Hepatic enzyme increased (Investigations) | 4 (4) | 1 (1)
Laboratory test abnormal (Investigations) | 2 (2) | 2 (2)
Blood insulin decreased (Investigations) | 0 (0) | 2 (2)
Blood pressure abnormal (Investigations) | 0 (0) | 1 (1)
Blood Thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Prothrombin time shortened (Investigations) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (18) | 9 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disk disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
gout (Metabolism and nutrition disorders) | 10 (25) | 15 (27)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 7 (7)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
No limitations or caveats are applicable to this summary

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data, information, inventions, discoveries, works, results, reports, presentations, intellectual property rights and whatever else arising out of the performance of the activities by PI, shall be of exclusive property of Sponsor or its designee(s). Sponsor shall be free to use the Results for publication or any other purpose, without any further obligations towards PI, and that, unless agreed in writing by Sponsor, PI shall have no right to publish, use or make presentations of the Results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT02500641/SAP_000.pdf
  • Study Protocol (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT02500641/Prot_001.pdf